CLINICAL TRIAL: NCT00880113
Title: The Dutch Acute Stroke Trial (DUST): Prediction of Outcome With CT-perfusion and CT-angiography
Brief Title: The Dutch Acute Stroke Trial (DUST): Prediction of Outcome With Computed Tomography (CT) - Perfusion and CT-angiography
Acronym: DUST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Dutch Heart Foundation (Other)
Responsible Party: B.K. Velthuis, University Medical Center Utrecht
Other Study IDs: 2008T034; NL25625.041.08
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Acute Stroke
Keywords: CT-perfusion; CT-angiography
MeSH Terms: conditions — Stroke | interventions — Cytidine Triphosphate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Acute stroke: Patients over 18 years of age with acute stroke symptoms of less then 9 hours duration and no hemorrhage on non-contrast CT.
  Interventions: Procedure: Non-contrast CT, CT-perfusion and CT-angiography

INTERVENTIONS:
Procedure: Non-contrast CT, CT-perfusion and CT-angiography — Included patients will undergo one additional combined CT-scan (NCCT, CTP and CTA) on day 3 (+/- 2 days).

SUMMARY:
Less than 10% of all ischemic stroke patients are treated by intravenous thrombolysis (IVT) as most present later than the accepted 3 hour time window. Intra-arterial thrombolysis (IAT) is possible 3-6 hours post ictus, but is infrequently used. Mechanical thrombectomy (MT) with a MERCI device is a new intervention possibility but lacks large randomized studies. Although it is desirable to treat more stroke patients, clinical information and plain CT alone are insufficient to discriminate which patients are most likely to benefit or be harmed from treatment. Advanced imaging techniques can help predict patient outcome and provide the necessary information to weigh expected benefit against associated risk of treatment. Visualizing the penumbra, the hypoperfused tissue at risk of infarction around the irreversible infarct core, is one way of identifying patients most likely to benefit from intervention. Magnetic resonance imaging (MRI) based selection of patients with sufficient penumbra for thrombolysis is possible, however, MR has less 24-hour availability than CT in the acute setting. Plain CT is mostly used to exclude intracerebral hemorrhage, and can easily be extended with CT perfusion (CTP) and CT angiography (CTA). CTP compares well to MRI for imaging penumbra and infarct core, and it is faster and more feasible than MRI. Other image findings such as infarct core size and leakage of the blood-brain-barrier (permeability) on CTP, and site and extent of the occlusion and collateral circulation on CTA also influence stroke outcome but have not been combined in one study to assess their combined predictive value.

Hypothesis:

The investigators hypothesize that combined CTP and CTA parameters can predict patient outcome in acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Acute neurological deficit caused by cerebral ischaemia
* Admission < 9 hours after onset of neurological deficit
* NIH Stroke Scale (NIHSS) of at least 2
* No absolute contraindications against intravenous contrast
* Informed consent from patient or family after admission scan
* Patients who awaken with stroke symptoms can only be included if they went to sleep without any stroke symptoms and the time from going to sleep until imaging is less than 9 hours

Exclusion Criteria:

* Neurological deficit caused by another diagnosis than cerebral ischaemia (such as intracerebral hemorrhage, subarachnoid hemorrhage or tumor)
* Patients with known contrast allergy or kidney failure
* Patients with the known combination of renal insufficiency and heart failure (New York Heart Association (NYHA) IV) will be excluded for the CTP and CTA scan at 3 days; they will have a non-contrast CT (NCCT) at that time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older with acute stroke symptoms who present in the hospital within 9 hours of onset of symptoms.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2009-05; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale | 90 days

SECONDARY OUTCOMES:
Final infarct size on CT | Day 3
Recanalization (CTA) | Day 3
Symptomatic hemorrhage | Day 3
Asymptomatic hemorrhage | Day 3

CONTACTS AND LOCATIONS:
Locations (14):
- Netherlands (14):
  - Academic Medical Center, Amsterdam
  - Onze Lieve Vrouwe Gasthuis (OLVG), Amsterdam
  - VU Medical Center, Amsterdam
  - Gelre Hospitals, Apeldoorn
  - Alysis Zorggroep, Arnhem
  - Catharina Hospital, Eindhoven
  - Leiden University Medical Center, Leiden
  - St. Antonius Hospital, Nieuwegein
  - UMC St. Radboud, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - St. Franciscus Gasthuis, Rotterdam
  - Medical Center Haaglanden, location Westeinde, The Hague
  - St. Elisabeth Hospital, Tilburg
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] Dankbaar JW, Horsch AD, van den Hoven AF, Kappelle LJ, van der Schaaf IC, van Seeters T, Velthuis BK; DUST Investigators. Prediction of Clinical Outcome After Acute Ischemic Stroke: The Value of Repeated Noncontrast Computed Tomography, Computed Tomographic Angiography, and Computed Tomographic Perfusion. Stroke. 2017 Sep;48(9):2593-2596. doi: 10.1161/STROKEAHA.117.017835. Epub 2017 Jul 17. PMID 28716981
- [Derived] Luitse MJ, Velthuis BK, Kappelle LJ, van der Graaf Y, Biessels GJ; DUST Study Group. Chronic hyperglycemia is related to poor functional outcome after acute ischemic stroke. Int J Stroke. 2017 Feb;12(2):180-186. doi: 10.1177/1747493016676619. Epub 2016 Oct 26. PMID 27784821
- [Derived] van den Wijngaard IR, Wermer MJ, Boiten J, Algra A, Holswilder G, Meijer FJ, Dippel DW, Velthuis BK, Majoie CB, van Walderveen MA. Cortical Venous Filling on Dynamic Computed Tomographic Angiography: A Novel Predictor of Clinical Outcome in Patients With Acute Middle Cerebral Artery Stroke. Stroke. 2016 Mar;47(3):762-7. doi: 10.1161/STROKEAHA.115.012279. Epub 2016 Jan 26. PMID 26814234
- [Derived] van den Wijngaard IR, Boiten J, Holswilder G, Algra A, Dippel DW, Velthuis BK, Wermer MJ, van Walderveen MA. Impact of Collateral Status Evaluated by Dynamic Computed Tomographic Angiography on Clinical Outcome in Patients With Ischemic Stroke. Stroke. 2015 Dec;46(12):3398-404. doi: 10.1161/STROKEAHA.115.010354. Epub 2015 Nov 5. PMID 26542691
- [Derived] Bennink E, Oosterbroek J, Horsch AD, Dankbaar JW, Velthuis BK, Viergever MA, de Jong HW. Influence of Thin Slice Reconstruction on CT Brain Perfusion Analysis. PLoS One. 2015 Sep 11;10(9):e0137766. doi: 10.1371/journal.pone.0137766. eCollection 2015. PMID 26361391
- [Derived] Luitse MJ, Velthuis BK, Dauwan M, Dankbaar JW, Biessels GJ, Kappelle LJ; Dutch Acute Stroke Study Group. Residual high-grade stenosis after recanalization of extracranial carotid occlusion in acute ischemic stroke. Stroke. 2015 Jan;46(1):12-5. doi: 10.1161/STROKEAHA.114.007169. Epub 2014 Dec 9. PMID 25492908
- [Derived] Fahmi F, Marquering HA, Borst J, Streekstra GJ, Beenen LF, Niesten JM, Velthuis BK, Majoie CB, vanBavel E; DUST study. 3D movement correction of CT brain perfusion image data of patients with acute ischemic stroke. Neuroradiology. 2014 Jun;56(6):445-52. doi: 10.1007/s00234-014-1358-7. Epub 2014 Apr 9. PMID 24715201